CLINICAL TRIAL: NCT03379987
Title: Analgesic Efficacy of Paravertebral Morphine for Acute Postoperative Pain: Randomized Multicenter Clinical Trial
Brief Title: Analgesic Efficacy of Paravertebral Morphine
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Diab Fuad Hetta, anesthesia and pain management departmewnt, SECI, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SECI-IRB-IORG0006563-404
Record Dates: First submitted 2017-12-17; First posted 2017-12-20 (Actual); Last update posted 2019-02-11 (Actual); Status verified 2019-02

CONDITIONS: Acute Pain
MeSH Terms: conditions — Acute Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PVB morphine (Experimental)
  Interventions: Drug: PVB morphine
- PVB bupivacaine (Active Comparator)
  Interventions: Drug: PVB bupivacaine

INTERVENTIONS:
Drug: PVB morphine — The PVB was performed under ultrasonographic guidance in the sitting position. Surgical disinfection of thoracoabdominal paravertebral area was done. A linear high-frequency transducer (10-12 MHz, Sonosite, Bothell, WA, USA) was used. The scanning process (Longitudinal out-of-plane technique) was started at 5-10 cm lateral to the spinous process of thoracic vertebrae to identify the rounded ribs and parietal pleura underneath. The transducer is then moved progressively more medially until the transverse processes are identified as more squared structure deeper to the ribs. A 100 mm needle was inserted out-of-plane to contact the transverse process of thoracic vertebra and then, walked off above the transverse process 1-1.5 cm deeper searching for loss of resistance injecting 10 ml of 0.25% bupivacaine + 3 mg morphine for group PVB morphine in incremental doses of 3 ml.
  Arms: PVB morphine
Drug: PVB bupivacaine — the same steps mentioned in group PVB morphine but the solution used for paravertebral block contain bupivacaine only 10 ml of 0.25% bupivacaine injected in in incremental doses of 3 ml.
  Arms: PVB bupivacaine

SUMMARY:
The investigator will test the analgesic efficacy of paravertebral morphine as an adjuvant to local anesthetics for acute postoperative pain following breast surgery and renal surgery

ELIGIBILITY:
Inclusion criteria

* Adult patients subjected to mastectomy or renal surgery

Exclusion criteria

* Patients complaining of coagulopathies
* Patients with vertebral anomalies

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-07 (Estimated); Study Completion 2019-08 (Estimated)

PRIMARY OUTCOMES:
24 hour postoperative morphine consumption | the first postoperative 24 hour
  the quantity of analgesic (morphine) consumed by the patient in the first postoperative 24 hour

SECONDARY OUTCOMES:
VAS pain score (visual analogue pain score) | we will assess every 4 hour in the first postoperative 24 hour
  a scle in which 0 = no pain and 10 = maximum tolerable pain

CONTACTS AND LOCATIONS:
Locations (1):
- Diab, Asyut, Assuit, Egypt